CLINICAL TRIAL: NCT03066362
Title: Respiratory Variations of the Inferior Vena Cava and Femoral Artery Flow to Predict Fluid Responsiveness in Spontaneously Breathing Patients With Sepsis, Acute Circulatory Failure, and Regular Cardiac Rhythm
Brief Title: Respiratory Variations for Predicting Fluid Responsiveness
Acronym: ReVaPreF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011_10; 2011-A00990-41 (Other: ID-RCB number)
Record Dates: First submitted 2016-11-09; First posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Sepsis; Respiratory Physiological Phenomena; Circulatory Failure
Keywords: Spontaneous ventilation
MeSH Terms: conditions — Sepsis; Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Echocardiography-Doppler (Experimental): Ultrasonographic recordings, systemic arterial pressure, heart rate, and respiratory rate are recorded immediately before and after volume expansion (VE), performed as a 30-minute infusion of 500 mL of 4% gelatin. Inferior Vena Cava diameters are measured during spontaneous and standardized respiratory cycles. Stroke volume is measured during spontaneous respiratory cycles.
  Interventions: Other: Echocardiography-Doppler

INTERVENTIONS:
Other: Echocardiography-Doppler — Ultrasonographic recordings are recorded immediately before and after volume expansion (VE), performed as a 30-minute infusion of 500 mL of 4% gelatin. Inferior Vena Cava diameters are measured during spontaneous and standardized respiratory cycles. Stroke volume is measured during spontaneous respiratory cycles.

SUMMARY:
Hypovolemia and acute circulatory failure affects more than 60% of patients hospitalized in intensive care or resuscitation. The volume expansion (VE) by fluid replacement therapy is the first treatment improve circulatory function. However, too much VE can be harmful. So, the use of dynamic predictive indicators of fluid responsiveness is recommended in patients with sepsis.In patients with spontaneous ventilation, few studies have evaluated these parameters. In mechanical ventilation, indices based on the respiratory variation of the diameters of vena cava have been studied and validated to predict the response to VE. However there is no similar study in spontaneously breathing patients without ventilatory support. The investigators hypothesize that the respiratory variations in the IVC diameters and femoral artery flow during standardized respiratory cycles are predictive factors of fluid responsiveness in spontaneously breathing patients with sepsis, acute circulatory failure, and regular cardiac rhythm.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of the intensive care units of the Lille university-hospital and of the Valenciennes general hospital.
* Age greater than or equal to 18.
* Patient insured
* Spontaneous breathing without ventilatory support or intubation or tracheotomy.
* Regular cardiac rhythm
* Prescription by the physician in charge of the patients of a 500 mL volume expansion in less than 30 minutes.
* Patients with sepsis with at least one sign of acute circulatory failure:

  * Tachycardia with heart rate> 100/min
  * systolic blood pressure <90mmHg or a decrease >40mmHg in previously hypertense patient
  * Oliguria <0.5ml/kg/hour for at least one hour
  * skin mottling

Exclusion Criteria:

* high-grade aortic insufficiency
* transthoracic echogenicity unsuitable for measuring the stroke volume or inferior vena cava diameters
* clinical signs of active exhalation
* clinical or ultrasonographic evidence of pulmonary edema due to heart failure
* pregnancy
* abdominal compartment syndrome
* Irregular cardiac rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-11; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
"respiratory variations in inferior vena cava diameters" with respect to the response to fluid resuscitation, assessed by the area under the ROC curve | during 30 minutes of the volume expansion

SECONDARY OUTCOMES:
"respiratory variations the femoral artery flow" with respect to the response to fluid resuscitation, assessed by the area under the ROC curve | during 30 minutes of the volume expansion

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Preau, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Intensive Care Department, Salengro Hospital, CHU de Lille, Lille, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No